CLINICAL TRIAL: NCT00354991
Title: An Open Label Study to Assess the Efficacy of Losartan/HCTZ Combination Therapy in Patients With Essential Hypertension Who Were Inadequately Controlled on Current Antihypertensive Monotherapy
Brief Title: Hyzaar Asia HEAALTH (0954A-950)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-950; MK0954A-950; 2006_012
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination

ARMS (1):
- 1 (Experimental): Losartan/HCTZ
  Interventions: Drug: losartan potassium (+) hydrochlorothiazide

INTERVENTIONS:
Drug: losartan potassium (+) hydrochlorothiazide — Patients took losartan 50 mg /HCTZ 12.5 mg orally once daily for 13 weeks. At Weeks 0, 4 and 8 if the blood pressure goal was not reached then the losartan/HCTZ combination will be titrated upwards according to the following scheme: losartan 50/HCTZ 12.5 to losartan 100/HCTZ 12.5 to losartan 100/HCTZ 25.

SUMMARY:
The objective of the study is to estimate the percentage of patients who reach blood pressure goal after 8 weeks of treatment with losartan/HCTZ combination.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and = 18 years of age
* Patients with essential hypertension previously treated with antihypertensive medications for at least 4 weeks but did not reach the blood pressure goal

Exclusion Criteria:

* History of any condition, therapy, lab abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient/subject to participate
* Pregnant or breastfeeding, or expecting to conceive within the projected duration of the study
* Previous history of severe essential hypertension
* History of stroke or myocardial infarction (heart attack)
* Evidence of renal or liver disease
* Uncontrolled diabetes mellitus
* Any known bleeding disorder
* Known sensitivity or intolerance to the study medication (losartan or hydrochlorothiazide)
* Other antihypertensive medications or medications that may affect blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2007-04-01 (Actual); Study Completion 2007-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching a blood pressure goal (diastolic <90mm Hg for non-diabetics; <80mm Hg for diabetics) after 8 weeks of treatment | 8 Weeks

SECONDARY OUTCOMES:
Safety and tolerability | 13 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Kim KS, Fan WH, Kim YD, Zhu W, Ngau YY, Tong P, Kim BS, Santos M, Lin WH, Buranakitjaroen P, Massaad R, Smith RD; Asia HEAALTH Study Investigators. Effectiveness of open-label losartan/hydrochlorothiazide combination therapy in Asian patients with hypertension not controlled with ACE inhibitor or ARB monotherapy. Hypertens Res. 2009 Jun;32(6):520-6. doi: 10.1038/hr.2009.42. Epub 2009 Apr 24. PMID 19390542
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html